CLINICAL TRIAL: NCT01282931
Title: Development and Implementation of a Patient-reported Outcome Questionnaire to Assess the Value of Progression-free Survival for Women With Metastatic Breast Cancer.
Brief Title: Patient-reported Outcome Questionnaire for Women With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Health Outcomes Solutions (Other)
Responsible Party: Principal Investigator, Susan Mathias, Principal Investigator, Health Outcomes Solutions
Other Study IDs: HOS-10-002
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Women; Stage IV; Metastatic; Breast Cancer; Progressed; Progression
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to understand the meaning of progression-free survival for women with metastatic breast cancer and to use this understanding to create and distribute a new questionnaire to assess the effect progression has on a woman's functioning and well-being.

DETAILED DESCRIPTION:
This study is being conducted in three stages. Stages I and II are complete. Participation in Stage III requires the completion of an online survey. The survey may be accessed at the following link:

https://www.surveymonkey.com/s/mbc3survey

Compensation options for eligible participants are listed at the end of the survey.

Eligibility will be confirmed in follow-up call/email by study staff.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 and older
* Clinical diagnosis of metastatic breast cancer
* U.S. resident
* Able to speak and read English
* Willing to sign and informed consent
* Willing to self-administer one online questionnaire that will take approximately 15 minutes to complete

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female 18 and older U.S. resident Clinical diagnosis of metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan D. Mathias, Principal Investigator — Health Outcomes Solutions
Locations (1):
- Health Outcomes Solutions, Winter Park, Florida, United States

REFERENCES:
- See also: Online location of study questionnaire — https://www.surveymonkey.com/s/mbc3survey